CLINICAL TRIAL: NCT00483626
Title: Hemodynamic Evaluation of Patients With Pulmonary Arterial Hypertension. Response to Sildenafil Treatment
Brief Title: Hemodynamic Response After Six Months of Sildenafil
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thorax-001-2003
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2007-06-07 (Estimated); Status verified 2007-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: hemodynamic; pulmonary hypertension; sildenafil
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oral sildenafil

SUMMARY:
The purpose of this study is to determine the clinical, functional and hemodynamic response after six months of sildenafil 50 mg TID in patients with pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension is a chronic devastating disease. There are few approval oral treatments. Sildenafil, a phosphodiesterase 5 inhibitors, has been recently approved for patients on functional class II and III showing hemodynamic benefits after 12 weeks of treatment. Long term hemodynamic evaluation after sildenafil treatment has not been evaluating in pulmonary arterial patients on functional class II to IV.

The protocol has been designed to evaluate patients on functional class II to IV from baseline conditions and after 6 months of sildenafil treatment (50 mg po TID). Clinical (functional class), functional (walked distance-6 minute walking test) and Hemodynamic evaluation is planned to be performed at baseline and after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 15 years old with Pulmonary arterial hypertension according with WHO hemodynamic definition,
* Who signed informed consent,
* Able to swallow tablets and follow instructions.

Exclusion Criteria:

* Patients with pulmonary hypertension with other categories than pulmonary arterial hypertension (associated to COPD, lund diseases, sleep apnea, thromboembolic disease, hight altitude), patients asymptomatic, patients who were responders to adenosine during hemodynamic test, patients treated with specific treatments for pulmonary arterial hypertension before started the study such as sildenafil, prostanoids, endothelin receptors blockers.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2003-08; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Arterial pulmonary resistance index | 6 months

SECONDARY OUTCOMES:
Mean pulmonary arterial pressure, Cardiac index, pulmonary saturation, walked distance, functional class. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Monica M Zagolin, MD, Principal Investigator — National Institute of Thorax
Locations (1):
- National Instiute of Thorax, Santiago, Metropolitanta, Chile

REFERENCES:
- [Background] Galie N, Ghofrani HA, Torbicki A, Barst RJ, Rubin LJ, Badesch D, Fleming T, Parpia T, Burgess G, Branzi A, Grimminger F, Kurzyna M, Simonneau G; Sildenafil Use in Pulmonary Arterial Hypertension (SUPER) Study Group. Sildenafil citrate therapy for pulmonary arterial hypertension. N Engl J Med. 2005 Nov 17;353(20):2148-57. doi: 10.1056/NEJMoa050010. PMID 16291984